CLINICAL TRIAL: NCT01518907
Title: A Phase 1b, Open-label, Dose-escalation Study of the Safety, Effectiveness, and Pharmacokinetics of AA4500 for the Treatment of Edematous Fibrosclerotic Panniculopathy Commonly Known as Cellulite
Brief Title: The Safety, Effectiveness, and Pharmacokinetics of AA4500 for the Treatment of Edematous Fibrosclerotic Panniculopathy (Commonly Known as Cellulite)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-830
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
Keywords: cellulite; Xiaflex
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- AA4500 0.0029 mg in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.0145 mg in 5 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.0145 mg in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.0435 mg in 5 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.0435 mg in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.116 mg in 5 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.116 mg in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.232 mg in 5 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 at 0.232 in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.464 mg in 5 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- AA4500 0.464 mg in 1 mL (Experimental)
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM

INTERVENTIONS:
Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM — Subdermal dose
  Other Names: XIAFLEX; XIAPEX

SUMMARY:
This study will evaluate the safety, effectiveness, pharmacokinetics, and immunogenicity of AA4500 at increasing doses and concentrations in the treatment of adult women with cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Be a female and be ≥ 21 years of age and ≤ 60 years of age
* Have a skin type classification of I through V according to the Fitzpatrick scale
* Have EFP within the posterolateral thigh(s) and/or buttock(s) for at least 12 months before the screening visit
* Have a photonumeric cellulite severity scale (CSS) score of ≥ 7 representing moderate to severe cellulite severity within the right or left buttock or the right or left posterolateral thigh (selected quadrant)
* Have an area of EFP within the selected quadrant that is at least 8 cm x 10 cm (ie, target EFP area) and is suitable for treatment:

  * The target EFP area must be located on the posterolateral thigh or within the buttock and does not involve the gluteal fold
  * The target EFP area must be evident when the subject is standing, without the use of any manipulation such as skin pinching or muscle contraction (ie, CSS Classification E score of 2 or 3) at screening and before injection
* Have a Body Mass Index (BMI) between 20.0 and 33.0 kg/m2, and intends to maintain stable body weight throughout the duration of the study (a variation of ≤5% from baseline body weight is permitted)
* Be willing to refrain from using artificial tanning devices and lotions during the 2-week period before screening and throughout the duration of the study
* Be willing to apply sunscreen with sun protection factor (SPF) ≥15 to the selected quadrant before each exposure to the sun while participating in the study (ie, screening through Day 90)
* Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at screening
* Have a negative urine pregnancy test at screening and before injection of AA4500 and be using an effective contraception method (ie, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for the duration of the study, or be surgically sterile, or be a postmenopausal female (no menses for at least 1 year or hysterectomy)
* Be willing and able to cooperate with the requirements of the study including requirements during the confinement period and throughout the study
* Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee/Human Research Ethics Committee (IRB/IEC/HREC). The subject must also sign an authorization form to allow disclosure of her protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
* Be able to complete and understand the various rating instruments in English

Exclusion Criteria:

* Has any of the following conditions:

  * Thyroid disease, unless controlled with medication for ≥ 6 months
  * Uncontrolled diabetes mellitus, as determined by the investigator
  * Uncontrolled hypertension, as determined by the investigator
  * Vascular disorder (eg, phlebitis or varicose veins) in area to be treated
  * Lipedema or a lymphatic disorder
  * History of lower extremity thrombosis or post-thrombosis syndrome
  * Documented autoimmune disorder such as lupus erythematosus, rheumatoid arthritis
  * Inflammation or active infection in area to be treated
  * Cutaneous alteration in area to be treated
  * Rash, eczema, psoriasis, or skin cancer in the area to be treated
  * History of keloidal scarring or abnormal wound healing
  * Coagulation disorder; taking an anticoagulant (except for ≤ 150 mg aspirin daily) up to 7 days prior to injection day
  * Known active hepatitis B or C (history of hepatitis A is permitted)
  * Known immune deficiency disease or a positive test for human immunodeficiency virus (HIV)
  * Other significant conditions including body dysmorphic disorder, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
* Has used any of the following for the treatment of EFP on the legs or buttock or intends to use any of the following at any time during the study:

  * Liposuction at any time before injection of AA4500
  * Injections (eg, mesotherapy); radiofrequency device treatments; laser treatment; or surgery (including subcision) within 12 months before injection of AA4500
  * Endermologie or similar treatments within 6 months before injection of AA4500
  * Massage therapy within 3 months before injection of AA4500
  * Creams to prevent or mitigate EFP within 2 weeks before injection of AA4500
* Has a tattoo in the quadrant selected for treatment
* Is presently nursing a baby or providing breast milk for a baby
* Intends to become pregnant during the study
* Intends to initiate an intensive sport or exercise program during the study
* Has an unrealistic expectation for treatment outcome, as determined by the investigator
* Has a positive alcohol breath test and/or a positive urine drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, and/or propoxyphene at screening or Day -1
* Has received an investigational drug or treatment within 30 days before injection of AA4500
* Has a known systemic allergy to collagenase or any other excipient of AA4500
* Has received any collagenase treatments within 30 days before treatment
* Has, at any time, received AA4500

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Investigator global aesthetic improvement scale assessment of the target cellulite area | Day 90
Subject global aesthetic improvement scale assessment of the target cellulite area | Day 90
A responder analysis based on proportion of subjects with a ≥ 30% improvement from baseline in the absolute surface depth of the central dimple/depression based on 3D digital photography. | Day 90
Percent change from baseline in total absolute surface depth of the central dimple/depression based on 3D digital photography. | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Urdaneta, MD MPH, Study Director — Endo Pharmaceuticals
Locations (1):
- SNBL Clinical Pharmacology Center, Inc, Baltimore, Maryland, United States